CLINICAL TRIAL: NCT02311829
Title: Evaluation d'un Dispositif de Suivi téléphonique Sur la Qualité de Vie Dans Les Crises Psychogènes Non Epileptiques.
Brief Title: Evaluation of a Telephone Follow-up Procedure on the Quality of Life in Psychogenic Non-epileptic Seizures
Acronym: EDUQ-CPNE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Central Hospital, Nancy, France (Other)
Collaborators: Dr Coraline HINGRAY (Unknown); Pr Raymund SCHWAN (Unknown); Dr Vincent LAPREVOTE (Unknown); Dr Jean Pierre VIGNAL (Unknown); Pr Hervé VESPIGNANI (Unknown); Dr Anne THIRIAUX (Unknown); Dr Delphine RAUCHER CHENE (Unknown); Dr Martine LEMESLE (Unknown); Dr Benoît TROJAK (Unknown); Pr Edouard HIRSCH (Unknown); Pr Pierre Vidailhet (Unknown); Dr Dominique Mastelli (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2012-A01580-43
Record Dates: First submitted 2014-10-28; First posted 2014-12-08 (Estimated); Last update posted 2016-03-08 (Estimated); Status verified 2016-03

CONDITIONS: Psychogenic Non Epileptic Seizure
Keywords: Quality of life, PNES, Epilepsy,
MeSH Terms: conditions — Psychogenic Nonepileptic Seizures; Epilepsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Telephone follow-up device (DST) (Experimental): An external independent clinical psychologist is responsible for calling regular the patient included in DST-arm.
  Telephone follow-up device(DST) consists of telephone calls at 15 day, 2 month and then every 2 months until 12 months. The clinical psychologist is designed to inform the patient about its pathology, promote acceptance of diagnosis, support the patient in his approach to care encouraging psychiatric observation. The device does not replace psychiatric counseling recommended.
  Interventions: Other: Telephone follow-up device
- Group control ; usual care (No Intervention): - Usual care: After diagnosis of PNES: orientation psychiatric care or CMP liberal and meeting biannually with the neurologist
  - For patients in both groups: in addition, quotation questionnaires of quality of life and evaluation by a neuropsychologist biannual for 24 months after the appointment with the neurologist.

INTERVENTIONS:
Other: Telephone follow-up device — For patients in the DST group only: Phone calls by clinical psychologist at J 15 at 2, then every 2 months until M12.
  Arms: Telephone follow-up device (DST)

SUMMARY:
The goal of this study is to evaluate effectiveness of the phone follow-up method compared to the conventional filler taken one.

DETAILED DESCRIPTION:
This study is a multicenter, non-drug therapy and randomized research trial, comparing a group of patients integrating the phone monitoring device (DST group) to a control group where patients are cared for in the usual way.

Subject recruiting modalities:

The study population represents patients diagnosis, PNES confirmed by following by the video-EEG, recorded in a center of epilepsy and in different CHU and informed of the diagnosis of PNES in a standardized manner.

Patients were recruited during their hospitalization video-EEG is conducted in part of the diagnostic workup of drug-resistant epilepsies, or demonstrations paroxysmal undetermined which may prove to be PNES.

Usual care:

After diagnosis of PNES: orientation psychiatric care or CMP liberal and meeting biannual with the neurologist.

In the study:

* For patients in both groups: Management usual care and, in addition, quotation questionnaires of quality of life and evaluation by a neuropsychologist biannually for 24 months after the appointment with the neurologist.
* For patients in the DST group only: Phone calls by psychologist at J 15, at 2 months, then every 2 months until M12. The device telephone follow (DST) consists of telephone calls (D15, M2, then every 2 months until M12) of the patient by an external independent psychologist designed to inform the patient about its pathology, promote acceptance of diagnosis, support the patient in his approach to care encouraging psychiatric observation. The device does not replace psychiatric counseling recommended.

ELIGIBILITY:
Inclusion Criteria:

* Patient above 18 years old
* Affiliation to social security
* Evolution disorders for over three months with at least 3 psychogenic non-epileptic seizures spaced over 24 hours and less than two years
* Diagnosis of PNES (associated or not with epilepsy) or laid confirmed following a video-EEG examination
* Standardized announcement of the disease made by a neurologist participant / PHRC training
* Good understanding of the French language
* Patient consented to participate in the study

Exclusion Criteria:

* Acute psychiatric pathology at the time of inclusion warranting urgent hospitalization (acute suicidal risk, Table delusional ...)
* Progressive neurological pathology intercurrent susceptible to aggravation for the duration of the study (glioma, multiple sclerosis, dementia ...)
* A patient who can not physically comply with the six-monthly review at the discretion of the investigator (planned move ...)
* Simultaneous participation to another therapeutic intervention study during the first 12 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 136 (Estimated)
Dates: Start 2014-01; Primary Completion 2018-01 (Estimated); Study Completion 2018-01 (Estimated)

PRIMARY OUTCOMES:
Evolution of quality of life scores every 6 months (From 6 to 24 months) | 24 months
  The primary endpoint is the assessment of quality of life scores measured at 6, 12, 18 and 24 months after start of treatment (visit D0) by self-administered questionnaires of quality of life (SF-36 general questionnaire quality of life) and QOLIE 31 (specific questionnaire epilepsy).

SECONDARY OUTCOMES:
Frequency of non epileptic seizures per month | 24 months (average for 6 months)
  Seizures diaries follow
Severity of seizures | 24 months
  Duration, injuries, loss of urine and feces, fall, loss of consciousness and subjective control feel of the listed crisis between 0 and 10 on EVA scale crisis control feel.
Psychiatric symptomology scores | 24 months
  Questionnaires (DSM-IV, Beck 21, MADRS, HAMA, DES, SDQ-20, TAS 20, Brief COPE)
Percentage of programmed psychological consultation and actually honored in medical and psychological center | 24 months
  This percentage is collected in medical and psychological center or from liberal psychiatrist \ psychologist (collected with phone call)
Number of urgent consultations or unprogrammed and \ or unprogrammed | 24 months
  consultations ( SAMU, emergency, reanimation, unprogrammed neurological consultations).

CONTACTS AND LOCATIONS:
Overall Officials: Louis MAILLARD, PU-PH, HDR, Principal Investigator — Central Hospital, Nancy, France
Locations (4):
- France (4):
  - Chu Strasbourg, Strasbourg, Alsace
  - Chu Dijon, Dijon, Bourgogne-Franche-Comté
  - Chu Reims, Reims, Champagne Ardennes
  - Chu Nancy, Nancy, Lorraine

REFERENCES:
- [Background] LaFrance WC Jr, Alosco ML, Davis JD, Tremont G, Ryan CE, Keitner GI, Miller IW, Blum AS. Impact of family functioning on quality of life in patients with psychogenic nonepileptic seizures versus epilepsy. Epilepsia. 2011 Feb;52(2):292-300. doi: 10.1111/j.1528-1167.2010.02765.x. Epub 2011 Feb 7. PMID 21299547
- [Background] Duncan R, Razvi S, Mulhern S. Newly presenting psychogenic nonepileptic seizures: incidence, population characteristics, and early outcome from a prospective audit of a first seizure clinic. Epilepsy Behav. 2011 Feb;20(2):308-11. doi: 10.1016/j.yebeh.2010.10.022. Epub 2010 Dec 30. PMID 21195031
- [Background] Goldstein LH, Chalder T, Chigwedere C, Khondoker MR, Moriarty J, Toone BK, Mellers JD. Cognitive-behavioral therapy for psychogenic nonepileptic seizures: a pilot RCT. Neurology. 2010 Jun 15;74(24):1986-94. doi: 10.1212/WNL.0b013e3181e39658. PMID 20548043
- [Background] Hingray C, Maillard L, Hubsch C, Vignal JP, Bourgognon F, Laprevote V, Lerond J, Vespignani H, Schwan R. Psychogenic nonepileptic seizures: characterization of two distinct patient profiles on the basis of trauma history. Epilepsy Behav. 2011 Nov;22(3):532-6. doi: 10.1016/j.yebeh.2011.08.015. Epub 2011 Oct 1. PMID 21962755
- [Background] Howlett S, Grunewald RA, Khan A, Reuber M. Engagement in psychological treatment for functional neurological symptoms--Barriers and solutions. Psychotherapy (Chic). 2007 Sep;44(3):354-60. doi: 10.1037/0033-3204.44.3.354. PMID 22122261
- [Background] Hubsch C, Baumann C, Hingray C, Gospodaru N, Vignal JP, Vespignani H, Maillard L. Clinical classification of psychogenic non-epileptic seizures based on video-EEG analysis and automatic clustering. J Neurol Neurosurg Psychiatry. 2011 Sep;82(9):955-60. doi: 10.1136/jnnp.2010.235424. Epub 2011 May 10. PMID 21561887
- [Background] Jirsch JD, Ahmed SN, Maximova K, Gross DW. Recognition of psychogenic nonepileptic seizures diminishes acute care utilization. Epilepsy Behav. 2011 Oct;22(2):304-7. doi: 10.1016/j.yebeh.2011.06.031. Epub 2011 Aug 2. PMID 21813334
- [Background] Josien E. Crises non épileptiques. EMC neurologie. 2005 ;1-9.
- [Background] LaFrance WC Jr, Keitner GI, Papandonatos GD, Blum AS, Machan JT, Ryan CE, Miller IW. Pilot pharmacologic randomized controlled trial for psychogenic nonepileptic seizures. Neurology. 2010 Sep 28;75(13):1166-73. doi: 10.1212/WNL.0b013e3181f4d5a9. Epub 2010 Aug 25. PMID 20739647
- [Background] Lesser RP. Psychogenic seizures. Neurology. 1996 Jun;46(6):1499-507. doi: 10.1212/wnl.46.6.1499. No abstract available. PMID 8649537
- [Background] Martin RC, Gilliam FG, Kilgore M, Faught E, Kuzniecky R. Improved health care resource utilization following video-EEG-confirmed diagnosis of nonepileptic psychogenic seizures. Seizure. 1998 Oct;7(5):385-90. doi: 10.1016/s1059-1311(05)80007-x. PMID 9808114
- [Background] Mayor R, Howlett S, Grunewald R, Reuber M. Long-term outcome of brief augmented psychodynamic interpersonal therapy for psychogenic nonepileptic seizures: seizure control and health care utilization. Epilepsia. 2010 Jul;51(7):1169-76. doi: 10.1111/j.1528-1167.2010.02656.x. Epub 2010 Jun 18. PMID 20561022
- [Background] Strutt AM, Hill SW, Scott BM, Uber-Zak L, Fogel TG. Motivation, psychopathology, locus of control, and quality of life in women with epileptic and nonepileptic seizures. Epilepsy Behav. 2011 Oct;22(2):279-84. doi: 10.1016/j.yebeh.2011.06.020. Epub 2011 Jul 23. PMID 21788158
- [Background] Worsley C, Whitehead K, Kandler R, Reuber M. Illness perceptions of health care workers in relation to epileptic and psychogenic nonepileptic seizures. Epilepsy Behav. 2011 Apr;20(4):668-73. doi: 10.1016/j.yebeh.2011.01.029. Epub 2011 Mar 25. PMID 21440511
- [Result] Abubakr A, Kablinger A, Caldito G. Psychogenic seizures: clinical features and psychological analysis. Epilepsy Behav. 2003 Jun;4(3):241-5. doi: 10.1016/s1525-5050(03)00082-9. PMID 12791325
- [Result] Al Marzooqi SM, Baker GA, Reilly J, Salmon P. The perceived health status of people with psychologically derived non-epileptic attack disorder and epilepsy: a comparative study. Seizure. 2004 Mar;13(2):71-5. doi: 10.1016/s1059-1311(03)00158-4. PMID 15129833
- [Result] Benbadis SR. How many patients with pseudoseizures receive antiepileptic drugs prior to diagnosis? Eur Neurol. 1999;41(2):114-5. doi: 10.1159/000008015. No abstract available. PMID 10023117
- [Result] Benbadis SR. A spell in the epilepsy clinic and a history of "chronic pain" or "fibromyalgia" independently predict a diagnosis of psychogenic seizures. Epilepsy Behav. 2005 Mar;6(2):264-5. doi: 10.1016/j.yebeh.2004.12.007. PMID 15710315
- [Result] Bodde NM, Brooks JL, Baker GA, Boon PA, Hendriksen JG, Aldenkamp AP. Psychogenic non-epileptic seizures--diagnostic issues: a critical review. Clin Neurol Neurosurg. 2009 Jan;111(1):1-9. doi: 10.1016/j.clineuro.2008.09.028. Epub 2008 Nov 18. PMID 19019531
- [Result] Bodde NM, Brooks JL, Baker GA, Boon PA, Hendriksen JG, Mulder OG, Aldenkamp AP. Psychogenic non-epileptic seizures--definition, etiology, treatment and prognostic issues: a critical review. Seizure. 2009 Oct;18(8):543-53. doi: 10.1016/j.seizure.2009.06.006. Epub 2009 Aug 13. PMID 19682927
- [Result] Carton S, Thompson PJ, Duncan JS. Non-epileptic seizures: patients' understanding and reaction to the diagnosis and impact on outcome. Seizure. 2003 Jul;12(5):287-94. doi: 10.1016/s1059-1311(02)00290-x. PMID 12810341
- [Result] Cuthill FM, Espie CA. Sensitivity and specificity of procedures for the differential diagnosis of epileptic and non-epileptic seizures: a systematic review. Seizure. 2005 Jul;14(5):293-303. doi: 10.1016/j.seizure.2005.04.006. PMID 15878291
- [Result] Duncan R, Oto M. Psychogenic nonepileptic seizures in patients with learning disability: comparison with patients with no learning disability. Epilepsy Behav. 2008 Jan;12(1):183-6. doi: 10.1016/j.yebeh.2007.09.019. PMID 18086462
- [Result] Fiszman A, Alves-Leon SV, Nunes RG, D'Andrea I, Figueira I. Traumatic events and posttraumatic stress disorder in patients with psychogenic nonepileptic seizures: a critical review. Epilepsy Behav. 2004 Dec;5(6):818-25. doi: 10.1016/j.yebeh.2004.09.002. PMID 15582828
- [Result] Goldstein LH, Deale AC, Mitchell-O'Malley SJ, Toone BK, Mellers JD. An evaluation of cognitive behavioral therapy as a treatment for dissociative seizures: a pilot study. Cogn Behav Neurol. 2004 Mar;17(1):41-9. doi: 10.1097/00146965-200403000-00005. PMID 15209224
- [Result] Guillemin F. Primer: the fallacy of subgroup analysis. Nat Clin Pract Rheumatol. 2007 Jul;3(7):407-13. doi: 10.1038/ncprheum0528. PMID 17599075
- [Result] Hall-Patch L, Brown R, House A, Howlett S, Kemp S, Lawton G, Mayor R, Smith P, Reuber M; NEST collaborators. Acceptability and effectiveness of a strategy for the communication of the diagnosis of psychogenic nonepileptic seizures. Epilepsia. 2010 Jan;51(1):70-8. doi: 10.1111/j.1528-1167.2009.02099.x. Epub 2009 Apr 27. PMID 19453708
- [Result] Iriarte J, Parra J, Urrestarazu E, Kuyk J. Controversies in the diagnosis and management of psychogenic pseudoseizures. Epilepsy Behav. 2003 Jun;4(3):354-9. doi: 10.1016/s1525-5050(03)00113-6. PMID 12791342
- [Result] LaFrance WC Jr, Barry JJ. Update on treatments of psychological nonepileptic seizures. Epilepsy Behav. 2005 Nov;7(3):364-74. doi: 10.1016/j.yebeh.2005.07.010. Epub 2005 Sep 16. PMID 16150653
- [Result] LaFrance WC Jr, Miller IW, Ryan CE, Blum AS, Solomon DA, Kelley JE, Keitner GI. Cognitive behavioral therapy for psychogenic nonepileptic seizures. Epilepsy Behav. 2009 Apr;14(4):591-6. doi: 10.1016/j.yebeh.2009.02.016. Epub 2009 Feb 20. PMID 19233313
- [Result] LaFrance WC Jr, Alper K, Babcock D, Barry JJ, Benbadis S, Caplan R, Gates J, Jacobs M, Kanner A, Martin R, Rundhaugen L, Stewart R, Vert C; NES Treatment Workshop participants. Nonepileptic seizures treatment workshop summary. Epilepsy Behav. 2006 May;8(3):451-61. doi: 10.1016/j.yebeh.2006.02.004. Epub 2006 Mar 15. PMID 16540377
- [Result] LaFrance WC Jr, Syc S. Depression and symptoms affect quality of life in psychogenic nonepileptic seizures. Neurology. 2009 Aug 4;73(5):366-71. doi: 10.1212/WNL.0b013e3181b04c83. PMID 19652140
- [Result] LaFrance WC Jr, Blum AS, Miller IW, Ryan CE, Keitner GI. Methodological issues in conducting treatment trials for psychological nonepileptic seizures. J Neuropsychiatry Clin Neurosci. 2007 Fall;19(4):391-8. doi: 10.1176/jnp.2007.19.4.391. PMID 18070841
- [Result] LaFrance WC Jr, Devinsky O. The treatment of nonepileptic seizures: historical perspectives and future directions. Epilepsia. 2004;45 Suppl 2:15-21. doi: 10.1111/j.0013-9580.2004.452002.x. PMID 15186340
- [Result] Lawton G, Mayor RJ, Howlett S, Reuber M. Psychogenic nonepileptic seizures and health-related quality of life: the relationship with psychological distress and other physical symptoms. Epilepsy Behav. 2009 Jan;14(1):167-71. doi: 10.1016/j.yebeh.2008.09.029. Epub 2008 Nov 6. PMID 18930164
- [Result] Lesser RP. Treating psychogenic nonepileptic seizures: easier said than done. Ann Neurol. 2003 Mar;53(3):285-6. doi: 10.1002/ana.10542. No abstract available. PMID 12601694
- [Result] Mokleby K, Blomhoff S, Malt UF, Dahlstrom A, Tauboll E, Gjerstad L. Psychiatric comorbidity and hostility in patients with psychogenic nonepileptic seizures compared with somatoform disorders and healthy controls. Epilepsia. 2002 Feb;43(2):193-8. doi: 10.1046/j.1528-1157.2002.20901.x. PMID 11903468
- [Result] Mrabet H, Mrabet A, Zouari B, Ghachem R. Health-related quality of life of people with epilepsy compared with a general reference population: a Tunisian study. Epilepsia. 2004 Jul;45(7):838-43. doi: 10.1111/j.0013-9580.2004.56903.x. PMID 15230710
- [Result] Oto M, Conway P, McGonigal A, Russell AJ, Duncan R. Gender differences in psychogenic non-epileptic seizures. Seizure. 2005 Jan;14(1):33-9. doi: 10.1016/j.seizure.2004.02.008. PMID 15642498
- [Result] Oxman AD, Guyatt GH. A consumer's guide to subgroup analyses. Ann Intern Med. 1992 Jan 1;116(1):78-84. doi: 10.7326/0003-4819-116-1-78. PMID 1530753
- [Result] Patrick DL, Chiang YP. Measurement of health outcomes in treatment effectiveness evaluations: conceptual and methodological challenges. Med Care. 2000 Sep;38(9 Suppl):II14-25. doi: 10.1097/00005650-200009002-00005. PMID 10982087
- [Result] Patrick DL, Deyo RA. Generic and disease-specific measures in assessing health status and quality of life. Med Care. 1989 Mar;27(3 Suppl):S217-32. doi: 10.1097/00005650-198903001-00018. PMID 2646490
- [Result] Picot MC, Crespel A, Daures JP, Baldy-Moulinier M, El Hasnaoui A. Psychometric validation of the French version of the quality of life in epilepsy inventory (QOLIE-31): comparison with a generic health-related quality of life questionnaire. Epileptic Disord. 2004 Dec;6(4):275-85. PMID 15634625
- [Result] Racine AD, Alderman EM, Avner JR. Effect of telephone calls from primary care practices on follow-up visits after pediatric emergency department visits: evidence from the Pediatric Emergency Department Links to Primary Care (PEDLPC) randomized controlled trial. Arch Pediatr Adolesc Med. 2009 Jun;163(6):505-11. doi: 10.1001/archpediatrics.2009.45. PMID 19487605
- [Result] Ramachandran K, Husain N, Maikhuri R, Seth S, Vij A, Kumar M, Srivastava N, Prabhakaran D, Airan B, Reddy KS. Impact of a comprehensive telephone-based disease management programme on quality-of-life in patients with heart failure. Natl Med J India. 2007 Mar-Apr;20(2):67-73. PMID 17802984
- [Result] Reuber M, Fernandez G, Bauer J, Helmstaedter C, Elger CE. Diagnostic delay in psychogenic nonepileptic seizures. Neurology. 2002 Feb 12;58(3):493-5. doi: 10.1212/wnl.58.3.493. PMID 11839862
- [Result] Reuber M. Psychogenic nonepileptic seizures: answers and questions. Epilepsy Behav. 2008 May;12(4):622-35. doi: 10.1016/j.yebeh.2007.11.006. Epub 2007 Dec 27. PMID 18164250
- [Result] Reuber M, Howlett S, Khan A, Grunewald RA. Non-epileptic seizures and other functional neurological symptoms: predisposing, precipitating, and perpetuating factors. Psychosomatics. 2007 May-Jun;48(3):230-8. doi: 10.1176/appi.psy.48.3.230. PMID 17478592
- [Result] Reuber M, Mitchell AJ, Howlett S, Elger CE. Measuring outcome in psychogenic nonepileptic seizures: how relevant is seizure remission? Epilepsia. 2005 Nov;46(11):1788-95. doi: 10.1111/j.1528-1167.2005.00280.x. PMID 16302859
- [Result] Reuber M, Pukrop R, Mitchell AJ, Bauer J, Elger CE. Clinical significance of recurrent psychogenic nonepileptic seizure status. J Neurol. 2003 Nov;250(11):1355-62. doi: 10.1007/s00415-003-0224-z. PMID 14648153
- [Result] Rusch MD, Morris GL, Allen L, Lathrop L. Psychological Treatment of Nonepileptic Events. Epilepsy Behav. 2001 Jun;2(3):277-283. doi: 10.1006/ebeh.2001.0180. PMID 12609370
- [Result] Salonen P, Tarkka MT, Kellokumpu-Lehtinen PL, Astedt-Kurki P, Luukkaala T, Kaunonen M. Telephone intervention and quality of life in patients with breast cancer. Cancer Nurs. 2009 May-Jun;32(3):177-90; quiz 191-2. doi: 10.1097/NCC.0b013e31819b5b65. PMID 19295417
- [Result] Sharpe D, Faye C. Non-epileptic seizures and child sexual abuse: a critical review of the literature. Clin Psychol Rev. 2006 Dec;26(8):1020-40. doi: 10.1016/j.cpr.2005.11.011. Epub 2006 Feb 10. PMID 16472897
- [Result] Sigurdardottir KR, Olafsson E. Incidence of psychogenic seizures in adults: a population-based study in Iceland. Epilepsia. 1998 Jul;39(7):749-52. doi: 10.1111/j.1528-1157.1998.tb01161.x. PMID 9670904
- [Result] Szaflarski JP, Hughes C, Szaflarski M, Ficker DM, Cahill WT, Li M, Privitera MD. Quality of life in psychogenic nonepileptic seizures. Epilepsia. 2003 Feb;44(2):236-42. doi: 10.1046/j.1528-1157.2003.35302.x. PMID 12558580
- [Result] Szaflarski JP, Szaflarski M, Hughes C, Ficker DM, Cahill WT, Privitera MD. Psychopathology and quality of life: psychogenic non-epileptic seizures versus epilepsy. Med Sci Monit. 2003 Apr;9(4):CR113-8. PMID 12709668
- [Result] Testa MA, Simonson DC. Assessment of quality-of-life outcomes. N Engl J Med. 1996 Mar 28;334(13):835-40. doi: 10.1056/NEJM199603283341306. No abstract available. PMID 8596551
- [Result] Testa SM, Schefft BK, Szaflarski JP, Yeh HS, Privitera MD. Mood, personality, and health-related quality of life in epileptic and psychogenic seizure disorders. Epilepsia. 2007 May;48(5):973-82. doi: 10.1111/j.1528-1167.2006.00965.x. Epub 2007 Feb 5. PMID 17284298
- [Result] Vaiva G, Vaiva G, Ducrocq F, Meyer P, Mathieu D, Philippe A, Libersa C, Goudemand M. Effect of telephone contact on further suicide attempts in patients discharged from an emergency department: randomised controlled study. BMJ. 2006 May 27;332(7552):1241-5. doi: 10.1136/bmj.332.7552.1241. PMID 16735333
- [Result] Wagner AK, Gandek B, Aaronson NK, Acquadro C, Alonso J, Apolone G, Bullinger M, Bjorner J, Fukuhara S, Kaasa S, Leplege A, Sullivan M, Wood-Dauphinee S, Ware JE Jr. Cross-cultural comparisons of the content of SF-36 translations across 10 countries: results from the IQOLA Project. International Quality of Life Assessment. J Clin Epidemiol. 1998 Nov;51(11):925-32. doi: 10.1016/s0895-4356(98)00083-3. PMID 9817109
- [Result] Ware JE Jr, Gandek B. Overview of the SF-36 Health Survey and the International Quality of Life Assessment (IQOLA) Project. J Clin Epidemiol. 1998 Nov;51(11):903-12. doi: 10.1016/s0895-4356(98)00081-x. PMID 9817107
- [Result] Witgert ME, Wheless JW, Breier JI. Frequency of panic symptoms in psychogenic nonepileptic seizures. Epilepsy Behav. 2005 Mar;6(2):174-8. doi: 10.1016/j.yebeh.2004.11.005. PMID 15710300
- [Result] Zaroff CM, Myers L, Barr WB, Luciano D, Devinsky O. Group psychoeducation as treatment for psychological nonepileptic seizures. Epilepsy Behav. 2004 Aug;5(4):587-92. doi: 10.1016/j.yebeh.2004.03.005. PMID 15256198
- [Result] The World Health Organization Quality of Life assessment (WHOQOL): position paper from the World Health Organization. Soc Sci Med. 1995 Nov;41(10):1403-9. doi: 10.1016/0277-9536(95)00112-k. PMID 8560308